CLINICAL TRIAL: NCT05373407
Title: A Randomized Controlled Trial Examining the Impact of Low Versus Moderate-intensity Aerobic Training in Post-discharge COVID-19 Older Subjects
Brief Title: Low Versus Moderate-intensity Aerobic Training in Post-discharge COVID-19 Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Ahmed Abdelmoniem Ibrahim, Associate professor, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00000
Record Dates: First submitted 2022-05-12; First posted 2022-05-13 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: COVID-19; Aerobic Exercises; Elderly
MeSH Terms: conditions — COVID-19 | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moderate intensity aerobic training (Experimental): The exercises were conducted at a heart rate of 50-70% of maximum heart rate for 30 minutes. Exercises were included strengthening muscles groups (shoulder flexors, extensors, abductor's muscles, hip flexors, extensor muscles, knee flexors, extensor muscles, abdominal muscles, and back muscles).
  Interventions: Other: aerobic exercise
- low intensity aerobic training (Experimental): Exercises were performed at 40-50% of the maximum heart rate Starting by 15 minutes of Warm-up time included static stretching of upper and lower body muscles.
  After that, participants performed 30 minutes of low-intensity aerobic training exercises, which included 20 minutes on the treadmill, followed by 10 minutes of cooling down.
  A set of 5-10 exercises was performed by each muscle group, three sets per exercise were performed, and 10-15 repetitions per series were performed 4 days per week
  Interventions: Other: aerobic exercise

INTERVENTIONS:
Other: aerobic exercise — participants will perform different dosage of the same intervention, one group will perform moderate intensity and the other will perform low intensity aerobic training

SUMMARY:
The main purpose of this study is to compare the impact of low versus moderate-intensity aerobic training in post-COVID 19 older subjects.

On exercise adherence and changes in physical fitness, psychological status, and quality of life after a 10-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 60 - 80 years with
* diagnosis of post-COVID-19

Exclusion Criteria:

* • History of lower limb surgeries, fractures

  * Cardiac problems
  * Respiratory problems
  * Neurological problems
  * Systemic problems and any other contraindications for aerobic training

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Distance walked in the 6-min walk test (6 MWT) | 8 weeks
  The 6-min walk test (6 MWT) measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD). (ATS Statement: Guidelines for the Six-Minute Walk Test, Am J Respir Crit Care Med, 2002)
Post-Covid Functional Scale (PCFS) | 8 weeks
  This scale measures the functional state and Independence of patients after COVID-19 infection. The scale includes two items scored from 0-4 and 0-5. A high value indicates more restrictions in function and independence during daily life.

SECONDARY OUTCOMES:
Number of repetitions performed in a 1-min Sit-to-Stand (STS) test | 8 weeks
  All 1-min STS tests are performed according to a standardized protocol by trained study staff. A standard chair is used with a flat seat and no armrests, stabilized against a wall. Patients are asked to sit with their legs hip-width apart and flexed to 90°, with their hands stationary on the hips.
2. Anxiety and Depression evaluated by the HAMLITON ScAnxiety and Depressionale (HADS) | 8 weeks
  Anxiety and Depression evaluated by the HAMLITON ScAnxiety and Depressionale (HADS)
Quality of life SF-36 | 8 weeks
  The SF-36 SF was used to evaluate self-reported domains of health status. This questionnaire consists of 36 items compiled into 8 scalesThe SF-36 questionnaire was used to evaluate self-reported domains of health status (Ware and Sherbourne, 1992). This questionnaire consists of 36 items compiled into 8 scales: physical functioning (PF), role functioning/physical (RP), bodily pain (BP), general health (GH), vitality (VT), social funct

CONTACTS AND LOCATIONS:
Locations (1):
- Hail University Poly Clinic, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No